CLINICAL TRIAL: NCT02709798
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Effect of Shenfu Injection on Reperfusion Injury in Patients With Acute ST Segment Elevation Myocardial Infarction After Primary Percutaneous Coronary Intervention: A Pilot Trial
Brief Title: ShenFu Injection for Myocardial Protection in Patients With Acute ST Segment Elevation Myocardial Infarction
Acronym: SF-STEMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: China Resources Sanjiu Medical & Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shao-Ping Nie, MD, PhD, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D99-2015(043)-TCM-4
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Myocardial Infarction
Keywords: Shenfu Injection; Reperfusion Injury; Myocardial Protection; Percutaneous Coronary Intervention
MeSH Terms: conditions — Myocardial Infarction; Reperfusion Injury | interventions — Shen-Fu; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Shenfu Injection (Experimental): 80ml Shenfu Injection + 70ml 5% glucose injection), ivdrip, 30 minutes before PCI and 1-5 days (once a day) after PCI (6 times in total). Drug titration time should be no less than 30 minutes.
  Interventions: Drug: Shenfu Injection
- 5% Glucose Injection (Placebo Comparator): 150 ml 5% glucose injection, ivdrip, 30 minutes before PCI and 1-5 days (once a day) after PCI (6 times in total). Drug titration time should be no less than 30 minutes.
  Interventions: Drug: 5% Glucose Injection

INTERVENTIONS:
Drug: Shenfu Injection
  Other Names: Shenfu Zhusheye
  Arms: Shenfu Injection
Drug: 5% Glucose Injection
  Arms: 5% Glucose Injection

SUMMARY:
The purpose of this study is to evaluate whether perioperative use of Shenfu Injection could reduce myocardial injury (enzymatic infarct size and infarct volume according to cardiac magnetic resonance imaging) in patients with STEMI after primary PCI

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and <75 years;
2. First-time acute anterior STEMI;
3. The time from onset of ischemic symptom to the time of initial PCI balloon inflation ≤6 hours;
4. >0.1 mV ST segment elevation in at least two contiguous precordial leads according to electrocardiogram;
5. Scheduled for primary PCI;
6. The presence of left anterior descending branch (LAD) occlusion in proximal or middle segment with pre-PCI TIMI flow 0 or 1 according to baseline coronary angiogram;
7. Written informed consent.

Exclusion Criteria:

1. Hypertrophic cardiomyopathy, aortic valve stenosis and/or regurgitation, pericarditis, or myocarditis;
2. Cardiogenic shock, severe ventricular arrhythmia, serious heart failure (Killip class III and above) or mechanical complications;
3. Patients after cardiopulmonary resuscitation (CPR) (including cardioversion);
4. Patients who have already received thrombolytic therapy;
5. Prior myocardial infarction or coronary artery bypass surgery;
6. Known serious hepatic, renal, blood, respiratory, or neuropsychiatric diseases;
7. Malignant tumor, lymphoma, HIV-positive, or hepatitis;
8. Uncontrolled hypertension (systolic BP >160 mm Hg or a diastolic BP >100 mmHg on at least two consecutive readings);
9. Patients with active bleeding, major surgery or trauma within 3 months and cerebrovascular accident within 6 months;
10. History of anemia (hemoglobin<90g/L) or thrombocytopenia (thrombocyte<90×109/L);
11. Multi-vessel disease with non-culprit vessel intervention;
12. Breastfeeding, pregnant, or potentially fertile women;
13. Patients who have known to be allergic to Shenfu Injection or its components or patients with serious adverse effect;
14. Patients with potential contraindication to CMR;
15. Participation in other clinical trial in recent 3 months;
16. Patients who cannot complete this trial or comply with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Infarct size | immediately after admission (0 hour), and 6, 12, 18, 24, 48, and 72 hours after PCI, as well as 4±1days after PCI
  Infarct size was assessed by measuring the area under the curve (AUC) of creatine kinase isoenzyme (CK-MB) within 72 hours after PCI and by performing cardiac magnetic resonance (CMR) imaging at 4±1days after PCI.

SECONDARY OUTCOMES:
AUC of cardiac troponin I (cTnI) | immediately after admission (0 hour), and 6, 12, 18, 24, 48, and 72 hours after PCI
Peak value of CK-MB and cTnI | 72 hours after PCI
ST segment resolution (%) according to ECG | up to 24 hours after PCI
Left ventricular end-diastolic diameter (LVEDD), left ventricular end-systolic diameter (LVESD), and Left ventricular ejection fraction (LVEF) | up to 28 days after PCI
Main adverse cardiovascular and cerebrovascular events (MACCE, including death, non-fatal myocardial infarction, target vessel revascularization, stroke, new-onset severe heart failure, re-hospitalization for heart failure) | up to 28 days after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Wang X, Miao H, Yan Y, Guo R, Gong W, He Y, Wang H, Ma X, Nie S. Effect of Shenfu Injection on Reperfusion Injury in Patients Undergoing Primary Percutaneous Coronary Intervention for ST Segment Elevation Myocardial Infarction: A Pilot Randomized Clinical Trial. Front Cardiovasc Med. 2021 Dec 3;8:736526. doi: 10.3389/fcvm.2021.736526. eCollection 2021. PMID 34926601